CLINICAL TRIAL: NCT01826448
Title: A Phase 1b Open Label, Dose Escalation Study to Assess Safety, Pharmacokinetics, Pharmacodynamics, and Antitumor Activity of PLX3397 in Combination With Vemurafenib in V600-mutated BRAF Unresectable or Metastatic Melanoma
Brief Title: A Phase 1b Open Label, Dose Escalation Study of PLX3397 in Combination With Vemurafenib in V600-mutated BRAF Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: No activity was observed. BRAFi-naïve participants should have received triple combination treatment (including MEK inhibitor). Continuation was not justified.
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Plexxikon (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLX108-09
Record Dates: First submitted 2013-04-01; First posted 2013-04-08 (Estimated); Results first posted 2020-05-28 (Actual); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: V600-mutated BRAF Unresectable Melanoma; V600-mutated BRAF Metastatic Melanoma; Stage III or Stage IV Metastatic Melanoma That Has Not Been Previously Treated With a Selective BRAF Inhibitor
MeSH Terms: interventions — pexidartinib; Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose extension cohort (Experimental): Patients will take PLX3397 and vemurafenib at the recommended phase 2 dose. This will be determined by the tolerability and safety of these drugs in the previous 3 cohorts.
  Interventions: Drug: PLX3397; Drug: vemurafenib
- Cohort 3 (Experimental): Patients will take 1000mg/day of PLX3397 and 960mg BID of vemurafenib
  Interventions: Drug: PLX3397; Drug: vemurafenib
- Cohort 2 (Experimental): Patients will take 800mg/day of PLX3397 and 960mg BID of vemurafenib
  Interventions: Drug: PLX3397; Drug: vemurafenib
- Cohort 1 (Experimental): Patients will take 800mg/day of PLX3397 and 720mg BID of vemurafenib
  Interventions: Drug: PLX3397; Drug: vemurafenib

INTERVENTIONS:
Drug: PLX3397
Drug: vemurafenib
  Other Names: Zelboraf

SUMMARY:
The purpose of this research study is to test the safety of an investigational new drug called PLX3397 when used in combination with Vemurafenib (Zelboraf™) at different dose levels. Vemurafenib has been approved by the United States Food and Drug Administration (FDA)/European Medicines Agency (EMA) for the treatment of a specific category of unresectable or metastatic melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years old.
* Patients with histologically confirmed unresectable Stage III or Stage IV metastatic melanoma who have not been previously treated with a selective BRAF inhibitor.
* Presence of a BRAF V600 mutation in the tumor tissue using the cobas BRAF mutation assay or comparable standard of care methodology.
* Measurable disease per RECIST v. 1.1 criteria.
* ECOG performance status 0 or 1.

Exclusion Criteria:

* Radiation therapy within 14 days of C1D1.
* Investigational drug use within 28 days of C1D1.
* Patients with active CNS lesions are excluded (i.e., those with radiographically unstable, symptomatic lesions). However, patients treated with stereotactic therapy or surgery are eligible if they remain without evidence of disease progression in the brain for ≥3 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11-05 (Actual); Primary Completion 2014-09-22 (Actual); Study Completion 2014-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (4):
  - UCLA, Los Angeles, California
  - University of Colorado, Denver, Aurora, Colorado
  - Vanderbilt University, Nashville, Tennessee
  - Seattle Cancer Care Alliance, Seattle, Washington
- Institute Gustave Roussy, Paris, France
- University Hospital Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 13 participants who met all inclusion and none of the exclusion criteria were enrolled in the study.
Pre-assignment Details: This was an open-label, multicenter, Phase 1b, dose-escalation study, followed by an Extension Phase at the recommended Phase 2 dose (RP2D) of both drugs. During Dose-escalation (planned n=40), cohorts of 3 to 6 participants were enrolled to identify the RP2D of each agent to be administered to patients enrolled in the subsequent Extension Phase.
Groups:
- Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID: Participant who received 800 mg/day (400 twice daily [BID]) of PLX3397 and 720 mg BID of vemurafenib.
- Cohort 2; PLX3397 800 mg/Day + Vemurafenib 960 mg BID: Participants who received 800 mg/day (400 twice daily [BID]) of PLX3397 and 960 mg BID of vemurafenib.
Period: Overall Study
Arm/Group | Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID | Cohort 2; PLX3397 800 mg/Day + Vemurafenib 960 mg BID
Started | 4 | 9
Completed | 0 | 0
Not Completed | 4 | 9
Not completed — Adverse Event | 1 | 3
Not completed — Disease progression | 2 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — 2 active cancers | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID | Cohort 2; PLX3397 800 mg/Day + Vemurafenib 960 mg BID | Total
Number analyzed (Participants) | 4 | 9 | 13
Age, Continuous [Mean (Full Range); unit: years] | 42 [35 to 52] | 60.1 [44 to 71] | 54.5 [35 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 5
  Male | 3 | 5 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events Who Received PLX3397 in Combination With Vemurafenib in V600-mutated BRAF Melanoma
Time Frame: 1 year
Population: Adverse events (AEs) were assessed in the modified intent-to-treat population (mITT).
Measure: Number; unit: percentage of participants
Arm/Group | Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID | Cohort 2; PLX3397 800 mg/Day + Vemurafenib 960 mg BID
Number analyzed (Participants) | 4 | 9
percentage of participants
  Any primary system organ class | 100 | 100
  Any AE | 100 | 100
  AEs related to both PLX3397 and vemurafenib | 100 | 55.6
  AEs related to PLX3397 | 75 | 77.8
  AEs related vemurafenib | 25 | 77.8
  AEs leading to withdrawal from any study treatment | 25 | 44.4
  AEs considered as dose limiting toxicities | 25 | 33.3
  Serious adverse events | 0 | 44.4
  Serious adverse events related to study treatment | 0 | 22.2
  Adverse events leading to death | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (and serious AEs [SAEs]) were recorded from the time the participant received the first dose of study drug up to 28 days after the last dose, up to 1 year (mITT population).
Description: Other non-serious adverse events occurring in ≥ 9 participants by system organ class or ≥ 3 participants by preferred term are reported from the mITT population.
Groups:
- Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID: Participant who received 800 mg/day (400 twice daily [BID] of PLX3397 and 720 mg BID of vemurafenib.
Arm/Group | Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID | Cohort 2; PLX3397 800 mg/Day + Vemurafenib 960 mg BID
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/4 | 4/9
Other Adverse Events (participants affected / at risk) | 4/4 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID (N=4) | Cohort 2; PLX3397 800 mg/Day + Vemurafenib 960 mg BID (N=9)
Alanine aminotransferase increased (Investigations) | 0 | 2
Neutrophil count decreased (Investigations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cerebellar haemorrhage (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1; PLX3397 800 mg/Day + Vemurafenib 720 mg BID (N=4) | Cohort 2; PLX3397 800 mg/Day + Vemurafenib 960 mg BID (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Constipation (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3
Fatigue (General disorders) | 1 | 7
Pyrexia (General disorders) | 0 | 4
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 2 | 5
Blood alkaline phosphatase increased (Investigations) | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 3
Blood creatinine increased (Investigations) | 1 | 2
Lymphocyte count decreased (Investigations) | 2 | 1
Weight decreased (Investigations) | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3

LIMITATIONS AND CAVEATS:
This study was terminated due to business decision before the planned sample size was reached; therefore, the planned outcome measure cannot be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No